CLINICAL TRIAL: NCT00633750
Title: Phase II Trial of OSI-774 (Tarceva), a Human Epidermal Growth Factor (HER) (erbB, Also Known as Epidermal Growth Factor Receptor, EGFR) Tyrosine Kinase Inhibitor, in Treatment-Naïve Operable Breast Cancer
Brief Title: Erlotinib in Treating Patients With Breast Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carlos L. Arteaga, Professor of Medicine and Cancer Biology, Associate Director of Clinical Research, Director VICC Breast Program, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 0222; VU-VICC-BRE-0222; VU-VICC-020448; P50CA098131 (NIH); R01CA080195 (NIH)
Record Dates: First submitted 2008-03-11; First posted 2008-03-12 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Erlotinib Hydrochloride; Immunohistochemistry; Chromatography, Liquid; Liquid Chromatography-Mass Spectrometry; Mass Spectrometry; Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tarceva (Experimental)
  Interventions: Drug: erlotinib hydrochloride; Genetic: TUNEL assay; Genetic: protein expression analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: liquid chromatography; Other: mass spectrometry; Other: matrix-assisted laser desorption ionization mass spectrometry; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: erlotinib hydrochloride — Tarceva will be given orally at a dose of 150 mg/day for 5-14 days. Patients are to undergo surgical resection of their tumor within 24 hours of the last dose of Tarceva.
  Other Names: OSI-774; erlotonib
Genetic: TUNEL assay — Used to assess drug-induced changes in tumor cell proliferation and cell death in pre-therapy and surgical specimens
Genetic: protein expression analysis — Used to assess drug-induced changes in tumor cell proliferation and cell death in pre-therapy and surgical specimens
Other: immunohistochemistry staining method — Used to assess drug-induced changes in tumor cell proliferation and cell death in pre-therapy and surgical specimens
Other: laboratory biomarker analysis — Used to assess level of expression of genetic markers in pre-therapy and surgical specimens
Other: liquid chromatography — Used to determine blood plasma levels of Erlotinib on the day of surgery
  Other Names: (LC/MS)
Other: mass spectrometry — Used to determine blood plasma levels of Erlotinib on the day of surgery
  Other Names: (LC/MS)
Other: matrix-assisted laser desorption ionization mass spectrometry — After treatment and following surgery, intervention will be used to determine Tarceva levels in tissue
  Other Names: MALDI MS
Procedure: therapeutic conventional surgery — Surgical treatment will occur within 24-hours following completion of therapy.

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving erlotinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well erlotinib works in treating patients with breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the in situ antitumor effect of neoadjuvant erlotinib hydrochloride as measured by a reduction in Ki67 and/or an increase in terminal deoxynucleotidyl transferase-mediated deoxyuridine triphosphate-biotin nick end labeling (TUNEL)-positive tumor cells in patients with treatment-naive, operable breast cancer.

Secondary

* To identify a molecular profile, based on measurements of Estrogen Receptor (ER), Epidermal Growth Factor Receptor (EGFR), and a Human Epithelial Growth Factor Receptor-2(HER2), and protein expression profiles in patients with treatment-naïve, operable breast cancer that is responsive to erlotinib hydrochloride.
* To correlate tumor concentrations of erlotinib hydrochloride with serum levels immediately before surgery.

OUTLINE: This is a multi-center study.

Patients receive oral erlotinib hydrochloride once daily for 5-14 days. Patients then undergo surgical resection within 24 hours after the last dose of erlotinib hydrochloride.

Tumor tissue samples are collected at baseline and during surgery for correlative laboratory studies. Tissue samples are stained for ER, HER2, and EGFR levels, proliferation (Ki67), and apoptosis (TUNEL) by immunohistochemistry. Levels of erlotinib hydrochloride in tissue samples are measured by matrix-assisted laser desorption/ionization mass spectrometry. Blood samples are collected on the day of surgery. Levels of erlotinib hydrochloride in blood samples are measured by liquid chromatography/mass spectrometry.

Patients are followed within 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage I or II (T1 or T2, N0 or N1) invasive mammary carcinoma

  * Diagnosis may be made by fine needle aspiration cytology or core biopsy

    * A repeat core biopsy is not required for patients who have a paraffin embedded diagnostic core biopsy specimen available for immunohistochemical staining

Exclusion Criteria:

* Patients with locally advanced disease who are planning to undergo preoperative neoadjuvant therapy are not eligible*

  * Locally advanced disease includes any of the following:

    * Primary tumor ≥ 5 cm (T3)
    * Tumor of any size with direct extension to the chest wall or skin (T4a-c)
    * Inflammatory breast cancer (T4d)
    * Fixed axillary lymph node metastases (N2)
    * Metastasis to ipsilateral internal mammary node (N3) NOTE: *Patients with primary tumors ≥ 5 cm (T3) or tumors involving the chest wall or skin who are not candidates for preoperative chemotherapy or who decline preoperative chemotherapy are eligible
* Measurable residual tumor at the primary site

  * Measurable disease is defined as any mass that can be reproducibly measured by physical examination
* Planning to undergo surgical treatment with either segmental resection or total mastectomy
* Patients with a prior history of contralateral breast cancer are eligible if they have no evidence of recurrence of their initial primary breast cancer
* No locally recurrent breast cancer
* No evidence of distant metastatic disease (i.e., lung, liver, bone, or brain metastases)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* ANC ≥ 1,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN
* Serum glutamic oxaloacetic transminase (SGOT) and serum glutamic pyruvic transminase (SGPT) ≤ 1.5 times ULN
* Must be at least 18 years old
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious medical illness that, in the judgement of the treating physician, places the patient at high risk of operative mortality

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for this primary breast cancer
* At least 7 days since prior tamoxifen or raloxifene as a preventive agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos L. Arteaga, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (5):
- United States (5):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period = 8/28/2002 through 10/16/2007
Pre-assignment Details: 54 participants were initially consented for this study. Four were determined to be ineligible. Three participants withdrew from the study before beginning.
Groups:
- Tarceva: Tarceva given by mouth at a dose of 150 mg/day for 5-14 days. Participants are to undergo surgical resection of their tumor within 24 hours of the last dose of Tarceva.
Period: Overall Study
Arm/Group | Tarceva
Started | 47
Completed | 42
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Tarceva
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing in Situ Anti-tumor Effect of Tarceva
Description: In situ anti-tumor effect of Tarceva as measured by a minimum 75% reduction in Ki67 compared to pre-treatment tumor cells in patients with operable breast cancer.
Time Frame: 5-14 days
Population: Patients who received the study drug and who had available pre- and post-treatment tissue.
Measure: Number; unit: participants
Groups:
- Tarceva: Following a pre-treatment core breast biopsy, participants are given Tarceva at a dose of 150 mg/day by mouth for 5-14 days. Within 24 hours of their last dose of Tarceva, participants undergo a post-treatment resection of their tumor.
Arm/Group | Tarceva
Number analyzed (Participants) | 34
participants | 8

2. Secondary Outcome: Molecular Profile of Participants Who Are Responsive to Tarceva
Description: Determined by estrogen receptor status (ER) and human epidermal growth factor receptor 2 (HER2) status, which are measured by staining of 200-500 tumor cells and noting the number stained. Positive = > 10% of cell show staining, negative = < 10% of cells show staining
Time Frame: at 5-14 days
Population: Participants with available pre- and post-treatment tissue and who demonstrated a post-treatment decrease in Ki67 levels compared to their pre-treatment levels
Measure: Number; unit: participants
Groups:
- Tarceva: Following a pre-treatment core biopsy, participants are given Tarceva at a dose of 150 mg/day by mouth for 5-14 days. Within 24 hours of their last dose of Tarceva, participants undergo a post-treatment resection of their tumor.
Arm/Group | Tarceva
Number analyzed (Participants) | 8
participants
  Estrogen receptor positive | 6
  Estrogen receptor negative | 2
  HER-2 positive | 1
  HER-2 negative | 7

3. Secondary Outcome: Average Post-treatment Plasma Level of Erlotinib Hydrochloride
Description: Post-treatment plasma level in µmol/L of erlotinib hydrochloride
Time Frame: After last dose of Tarceva, at 5-14 days, and before surgery
Population: Participants with blood taken within 24 hours of last dose of erlotinib and before surgery
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- Tarceva: Following a pre-treatment core biopsy, participants are given Tarceva at a dose of 150 mg/day by mouth for 5-14 days. Within 24 hours of their last dose of Tarceva, participants have their blood drawn and then undergo surgical resection of their tumor.
Arm/Group | Tarceva
Number analyzed (Participants) | 30
µmol/L | 8.8 (7.4)

ADVERSE EVENTS:
Arm/Group | Tarceva
Serious Adverse Events (participants affected / at risk) | 1/47
Other Adverse Events (participants affected / at risk) | 44/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tarceva (N=47)
Pulmonary ebmolisim (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tarceva (N=47)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Alkaline phosphatase (Investigations) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 3 (3)
Arthiritis (Musculoskeletal and connective tissue disorders) | 9 (9)
Blurred vision (Eye disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 15 (15)
Fatigue (General disorders) | 9 (9)
Headache (Nervous system disorders) | 7 (7)
Hemoglobin (Investigations) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Hypertension (Vascular disorders) | 7 (7)
Hypothyroidism (Endocrine disorders) | 3 (3)
Infection (without neutropenia) (Infections and infestations) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Joint, muscle or bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Mood Changes - depression (Psychiatric disorders) | 3 (3)
Mood Changes-anxiety/agitation (Psychiatric disorders) | 11 (11)
Mucositis (Gastrointestinal disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (7)
Pain (General disorders) | 19 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11)
Rash (Skin and subcutaneous tissue disorders) | 29 (29)
SGPT (ALT) (Investigations) | 3 (3)
Hot flashes/flushes (Vascular disorders) | 7 (7)
High cholesterol (Investigations) | 5 (5)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes